CLINICAL TRIAL: NCT02852837
Title: A Phase 1, Open-label, Dose Escalation Study of JNJ-54767414 (Daratumumab) in Chinese Subjects With Relapsed or Refractory Multiple Myeloma Who Failed at Least 2 Prior Lines of Systemic Therapy
Brief Title: Dose Escalation Study of JNJ-54767414 (Daratumumab) in Chinese Participants With Relapsed or Refractory Multiple Myeloma Who Failed at Least 2 Prior Lines of Systemic Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108180; 54767414MMY1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: Dose Escalation Part (Experimental): Participants will receive single dose of daratumumab from Week 1 till Week 3 (Period 1 - single dosing period) followed by 6 weekly doses of daratumumab until Week 9 (Period 2 - weekly dosing period) and every 2 weeks for 8 infusions and then once every 4 weeks from Week 26 until disease progression, intolerability, or other reasons for treatment discontinuation (Period 3 - less intense dosing period). A dose of 8 milligram per kilogram (mg/kg) will be chosen as the starting dose and will be escalated to 16 mg/kg if the 8 mg/kg is determined safe and tolerated by study evaluation team (SET).
  Interventions: Drug: Daratumumab
- Part 2: Pharmacokinetic (PK) Expansion Part (Experimental): Participants will receive daratumumab at 16 mg/kg in 3 periods as given in the Part 1.
  Interventions: Drug: Daratumumab
- Part 3: Safety Expansion Part (Experimental): Participants will receive daratumumab 16 mg/kg every week for 8 weeks followed by every 2 weeks for an additional 16 weeks, and then every 4 weeks thereafter. Participants will be treated with daratumumab until disease progression, intolerability, or any other reasons for treatment discontinuation.
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — Intravenous (IV) infusion of 8 mg/kg or 16 mg/kg daratumumab.
  Other Names: JNJ-54767414

SUMMARY:
The purpose of this study is to evaluate the tolerability, safety and the pharmacokinetic (PK) profile of daratumumab in Chinese participants with relapsed or refractory multiple myeloma (RRMM) who failed at least 2 prior lines of systemic therapy (Part 1 and Part 2); and to evaluate the tolerability and safety of daratumumab in Chinese participants whose prior therapy included a proteasome inhibitor (PI) and an immunomodulatory drug (IMiD) and who have demonstrated disease progression on the last therapy (Part 3).

ELIGIBILITY:
Inclusion Criteria:

Part 1 and 2:

* Chinese participant who must be at least 20 years of age
* Documented multiple myeloma (MM) with measurable disease according to protocol-defined criteria
* Relapsed or refractory multiple myeloma after receiving at least 2 prior lines of therapy
* Eastern Cooperative Oncology Group performance status score of 0, 1, or 2
* Adequate recovery from prior therapy

Part 3:

* Chinese participants who must be at least 18 years of age
* Received both a proteasome inhibitor (PI) (greater than or equal to [>=] 2 cycles or 2 months of treatment) and an immunomodulatory drug (IMiD) (>=2 cycles or 2 months of treatment) in any order during the course of treatment (except for participants who discontinued either of these treatments due to a severe allergic reaction within the first 2 cycles/months)
* Documented evidence of progressive disease (PD) based on investigator's determination of response as defined by the International Myeloma Working Group (IMWG) criteria on or after their last regimen

Exclusion Criteria:

Part 1 and 2:

* Received daratumumab or other anti-CD38 therapies previously
* Previously received an allogenic stem cell transplant or has received an autologous stem cell transplantation within 12 weeks
* Exhibiting clinical signs of meningeal involvement of multiple myeloma
* Known chronic obstructive pulmonary disease, known moderate or severe persistent asthma within the past 2 years, or uncontrolled asthma of any classification
* Known clinically significant cardiac disease
* Known to be seropositive for human immunodeficiency virus, hepatitis B or known to have a history of hepatitis C
* Has plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), or amyloidosis
* Abnormal laboratory values according to protocol-defined parameters at screening

Part 3:

- Received anti-myeloma treatment within 2 weeks before Cycle 1, Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-09-26 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) as a Measure of Safety and Tolerability (Part 1,2 and 3) | From the time of signing of informed consent form (ICF) until 30 days after the last study drug dose (approximately 2 years)
Maximum Observed Plasma Concentration (Cmax) (Part 1 and 2) | Until Cycle 14, Day 1 (each cycle of 21 days till Cycle 3 and 28 days Cycle 4 onward)
  The Cmax is the maximum observed plasma concentration.
Trough Analyte Concentration (Ctrough) (Part 1 and 2) | Until Cycle 14, Day 1 (each cycle of 21 days till Cycle 3 and 28 days Cycle 4 onward)
  The (Ctrough) is the concentration before dosing just prior to the beginning of a doing interval.
Area Under the Plasma Concentration-Time Curve (AUC) (Part 1 and 2) | Until Cycle 14, Day 1 (each cycle of 21 days till Cycle 3 and 28 days Cycle 4 onward)
  AUC is defined as area under the plasma concentration-time curve.
Systemic Clearance (CL) (Part 1 and 2) | Until Cycle 14, Day 1 (each cycle of 21 days till Cycle 3 and 28 days Cycle 4 onward)
  Systemic Clearance (CL) is a quantitative measure of the rate at which a drug substance is removed from the body. The total systemic clearance after intravenous dose was estimated by dividing the total administered dose by the plasma Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]).
Elimination Half-Life (t1/2) (Part 1 and 2) | Until Cycle 14, Day 1 (each cycle of 21 days till Cycle 3 and 28 days Cycle 4 onward)
  Elimination half-life (t[1/2]) is associated with the terminal slope (lambda [z]) of the semi-logarithmic drug concentration-time curve, calculated as 0.693/lambda(z).
Volume of Distribution (Vd) (Part 1 and 2) | Until Cycle 14, Day 1 (each cycle of 21 days till Cycle 3 and 28 days Cycle 4 onward)
  The Vd is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | From the date of first dose of daratumumab to the date of initial documentation of progressive disease (approximately 2 years)
  ORR is defined as the proportion of participants who achieve complete response [CR] (including sCR) according to the IMWG criteria, during or after the study treatment. IMWG criteria CR: Negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas and less than (<)5 % plasma cells (PCs) in bone marrow; sCR: CR along with normal free light chain (FLC) ratio and absence of clonal PCs by immunohistochemistry, immunofluorescence or 2 to 4 color flow cytometry. Partial Response (PR): more than equal to (>=) 50percent (%) reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90% or to <200 mg/24 hours; VGPR: Serum and urine M-component detectable by immunofixation but not on electrophoresis, or >= 90 % reduction in serum M-protein plus urine M-protein less than (<)100 mg/24 hours.
Time to Response | From the date of first dose of daratumumab to the date of initial documentation of a response (approximately 2 years)
  Time to response is defined as the time between the date of first dosing and the first efficacy evaluation that the participant has met all criteria for PR (including VGPR) or CR (including sCR).
Duration of Response | From the date of initial documentation of a response to the date of first documented evidence of progressive disease (approximately 2 years)
  Duration of Response will be calculated from date of initial documentation of a response (CR/PR) to date of first documented evidence of PD. IMWG criteria for PD- Increase of 25% from lowest response value in any one of following: Serum M-component (absolute increase must be >=0.5 gram per deciliter [g/dL]), urine M-component (absolute increase must be >=200 mg/24 hours), only in participants without measurable serum and urine M-protein levels: difference between involved and uninvolved FLC levels (absolute increase must be >10 mg/dL), only in participants without measurable serum and urine M-protein levels and without measurable disease by FLC levels, bone marrow PC percentage (absolute percentage must be >=10%). Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in size of existing bone lesions or soft tissue plasmacytomas. Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed to PC proliferative disorder.
Progression-Free Survival (PFS) | From the date of first dose of daratumumab to the date of first documented progressive disease (approximately 2 years)
  PFS is defined as the time from the date of first dose of daratumumab to the date of first documented Progressive disease (PD), as per International Myeloma Working Group (IMWG) criteria, or death due to any cause, whichever occurs first.
Overall Survival (OS) | From the date of first dose of daratumumab to the date of the participant's death (approximately 2 years)
  Overall survival (OS) is measured from the date of first dose of daratumumab to the date of the participant's death.
Number of Participants With Incidence of Antibodies to Daratumumab | Up to Follow-up Phase-Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (5):
- China (5):
  - Beijing
  - Hangzhou
  - Shanghai
  - Suzhou
  - Tianjin

REFERENCES:
- [Derived] Li X, Dosne AG, Perez Ruixo C, Perez Ruixo JJ. Pharmacodynamic-Mediated Drug Disposition (PDMDD) Model of Daratumumab Monotherapy in Patients with Multiple Myeloma. Clin Pharmacokinet. 2023 May;62(5):761-777. doi: 10.1007/s40262-023-01232-8. Epub 2023 Apr 6. PMID 37022569
- [Derived] Jing H, Yang L, Qi J, Qiu L, Fu C, Li J, Yang M, Qi M, Fan N, Ji J, Lu J, Li Y, Jin J. Safety and efficacy of daratumumab in Chinese patients with relapsed or refractory multiple myeloma: a phase 1, dose-escalation study (MMY1003). Ann Hematol. 2022 Dec;101(12):2679-2690. doi: 10.1007/s00277-022-04951-3. Epub 2022 Oct 27. PMID 36301338
- See also: A Phase 1, Open-label, Dose Escalation Study of JNJ-54767414 (Daratumumab) in Chinese Subjects With Relapsed or Refractory Multiple Myeloma Who Failed at Least 2 Prior Lines of Systemic Therapy — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR108180&attachmentIdentifier=73dbcc08-6b56-4322-a2db-6ec64f3e2398&fileName=CR108180_CSR_Synopsis.pdf&versionIdentifier=